CLINICAL TRIAL: NCT02974335
Title: A Phased-Implementation Feasibility and Proof-of-Concept Study to Assess Incorporating the NIDA CTN Common Data Elements (CDEs) Into the Electronic Health Record (EHR) in Large Primary Care Settings ("CDE-EHR-PC" Study), Phase 1
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Oregon Health and Science University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01948
Record Dates: First submitted 2016-11-10; First posted 2016-11-28 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Care Providers (PCPs): Key stakeholders including: informatics/Epic leaders, medical providers, and patients from the two health systems that will be involved in the study, as well as national health information technology leaders from other large health systems.
  Interventions: Behavioral: Interviews with Stakeholders
- Medical Assistants (MAs) + Registered Nurses (RNs): Key stakeholders including: informatics/Epic leaders, medical providers, and patients from the two health systems that will be involved in the study, as well as national health information technology leaders from other large health systems.
  Interventions: Behavioral: Interviews with Stakeholders
- Patients: Key stakeholders including: informatics/Epic leaders, medical providers, and patients from the two health systems that will be involved in the study, as well as national health information technology leaders from other large health systems.
  Interventions: Behavioral: Interviews with Stakeholders

INTERVENTIONS:
Behavioral: Interviews with Stakeholders — The information gained from stakeholders will be applied in an iterative process to develop a best-practice approach to screening patients, and to build the EHR tools (CDEs and CDS) that will be further tailored and tested in Phase 2, and then implemented in one clinic in Phase 3.

SUMMARY:
This is a 4-phase study to implement the NIDA CDEs in primary care settings. Collecting and utilizing the CDEs in clinical practice requires a strategy for implementing screening to collect substance use information that populates the CDEs, and assisting primary care providers to offer appropriate interventions by providing clinical decision support (CDS) and a mechanism for making referrals to addiction treatment. We aim to maximize the efficient adoption of screening, CDS, and treatment referrals by integrating all of these activities into the electronic health record (EHR).

The study will be conducted at three sites, representing three large health systems. Each phase will include deliverables essential to move to the next phase, and an independent Advisory Committee will review progress and make recommendations at each transition about how best to progress to each subsequent phase. Based on progress during earlier phases, the Advisory Committee may recommend expansion to additional clinics or health systems during the second part of Phase 4.

DETAILED DESCRIPTION:
Phase 1 involves identifying the optimal screening tools and approaches for capturing CDE data, programming the screening tools and CDEs into the Epic EHR, and soliciting stakeholder input regarding implementation strategies for screening and clinical interventions (including treatment referrals) to address substance use.

In the KTA framework, Phase 1 addresses the first steps in the action cycle, which are to identify, review, and select the tools that are to be implemented; adapt tools to the local context; assess barriers to use of the tools; and begin the process of implementation by programming these tools into the Epic EHR. We will accomplish these steps primarily through interviews and focus groups with key stakeholders. The information gained from stakeholders will be applied in an iterative process to develop a best-practice approach to screening patients, and to build the EHR tools (CDEs and CDS) that will be further tailored and tested in Phase 2, and then implemented in one clinic in Phase 3.

Research Questions and Aims

The research questions that Phase 1 seeks to address are:

1. Where should screening and initial assessment occur, and who should administer the screening and assessment questionnaires?
2. Is it better to screen for drugs only, or for drugs and alcohol, or for drugs, alcohol and tobacco? Should screening also include depression (e.g., PHQ2 and PHQ9)? Should screening be embedded in a broad behavioral health screen (e.g., a comprehensive health risk assessment such as My Own Health Report (30))?

The specific aim that corresponds to Phase 1 is Aim 1: To program the NIDA CTN CDEs and a lean decision support module into Epic. This phase will also define potential barriers and facilitators to the adoption of the CDEs and CDS, which is a component of Specific Aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current primary care clinic patient

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the three clinics where we plan to implement study Phases 2-4. Clinic staff will give recruitment flyers to all patients registering for appointments in the week prior to each focus group. Potential participants who are interested in participating will call the Research Coordinator, who will assess eligibility and schedule them for the appropriate group. Groups will be divided based on age; one group will include participants under age 50, and a second group will include those age 50 and over. This grouping strategy is chosen because individuals in these age groups are anticipated to differ in their substance use patterns, medical needs, and concerns about screening procedures.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Patient level outcomes: diagnosis, and treatment referral | 1 Year
Provider level outcomes: screening and assessment, and clinical interventions including counseling and treatment referral. | 1 year
Systems level outcomes: logistics and costs of introducing the CDEs. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, Principal Investigator — New York University Medical School
Locations (3):
- United States (3):
  - Massachusettes General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Result] McNeely J, Kumar PC, Rieckmann T, Sedlander E, Farkas S, Chollak C, Kannry JL, Vega A, Waite EA, Peccoralo LA, Rosenthal RN, McCarty D, Rotrosen J. Barriers and facilitators affecting the implementation of substance use screening in primary care clinics: a qualitative study of patients, providers, and staff. Addict Sci Clin Pract. 2018 Apr 9;13(1):8. doi: 10.1186/s13722-018-0110-8. PMID 29628018